CLINICAL TRIAL: NCT00006062
Title: Phase I Study of Oxaliplatin in Patients With Advanced Malignancies and Varying Degrees of Liver Dysfunction
Brief Title: Oxaliplatin to Treat Advanced Cancers With Liver Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000172; 00-C-0172
Record Dates: First submitted 2000-07-11; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-06

CONDITIONS: Liver Disease
Keywords: Liver Impairment; Pharmacokinetics; Platinum Analogues
MeSH Terms: conditions — Liver Diseases | interventions — Oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
This is a phase I study of the experimental anticancer drug oxaliplatin. It is designed to establish the maximum dose of the drug that can be given safely to patients with cancer who have impaired liver function and to determine the drug's side effects. It will also examine how liver function affects the drug's elimination from the body. The liver plays an important role in the elimination of many anticancer drugs, and patients with impaired liver function should not take certain drugs or should take them in reduced doses.

Patients 18 years of age and older with cancer that has metastasized (spread from the original tumor site) and for whom standard treatment is not available or is no longer effective may be eligible for this study. Candidates will be screened with various tests and procedures that may include physical examination, computerized tomography (CT) or magnetic resonance imaging (MRI) scans, chest X-rays, and blood and urine tests.

Participants will be given oxaliplatin in doses determined according to their level of liver function. Patients may have normal liver function or mildly, moderately or severely impaired liver function, or may have had a liver transplant. Oxaliplatin will be infused intravenously (through a vein) over two hours on the first day of 21-day treatment cycles-that is, once every 3 weeks. Treatment will continue as long as the cancer is under control and side effects do not require stopping the drug. Urine will be collected over 48 hours after the infusion to determine how much of the drug is eliminated in urine. Blood tests will be done to monitor safety of the treatment, and imaging studies, such as X-rays, CT and MRI scans, will be done periodically to evaluate the tumor's response to treatment.

Special blood tests will also be done to study how oxaliplatin is eliminated from the body. With the first dose of the drug, blood samples will be collected just before the infusion begins, just before it ends, 15 minutes, 30 minutes, 1, 2, 4, 6, 24, 48, and 72 hours after the infusion, and again 1 week and 3 weeks later. Additional blood samples may be collected at the third treatment cycle.

DETAILED DESCRIPTION:
Oxaliplatin is a diaminocyclohexane platinum derivative with known anticancer activity in solid tumors. The recommended single-agent dose of oxaliplatin in adult cancer patients is 130 mg/m(2) given intravenously over 2 hours every 3 weeks. Hepatic metabolism is the major route of drug elimination for many anti-cancer agents. Although there is limited safety and pharmacokinetic data for oxaliplatin in patients with renal impairment, there is currently no data regarding its disposition in patients with liver dysfunction. This phase I and pharmacologic study of a single agent oxaliplatin is being conducted in adult cancer patients with advanced malignancies and varying degrees of liver dysfunction. Patients will be stratified into five groups based upon their degree of liver dysfunction as assessed by liver function tests. Group A will consist of patients with normal hepatic function to serve as pharmacologic controls. Group E will consist of patients who have received a liver transplant. The remaining 3 groups will start at different doses of oxaliplatin based on hepatic dysfunction and dose escalation in these groups will proceed in a manner in accordance with standard phase I trial with 3 patients per dose level until dose limiting toxicity is observed. Pharmacokinetic monitoring will be performed in all patients on study. The goals of this trial are to define the toxicities and pharmacokinetics of single agent oxaliplatin in this patient population and to determine recommended doses of oxaliplatin in patients with different degrees of hepatic impairment.

ELIGIBILITY:
Must have histologically confirmed malignancy which is metastatic or unresectable and for which standard curative or palliative treatments do not exist or are no longer effective.

Must have had 3 or fewer previous regimens (may have included prior platinum therapy). Previous radiation allowed but should have included less than or equal to 30% of bone marrow.

At least 18 years old.

Karnofsky performance status greater than or equal to 60%. Patients should have an expected survival of at least 2 months.

Leukocytes greater than or equal to 3,000/micro liter; or absolute neutrophil count greater than or equal to 1,500/micro liter; or platelets greater than or equal to 100,000/micro liter, creatinine within normal institutional limits; or measured creatinine clearance greater than or equal to 60 mL/min for patients with creatinine levels above institutional normal.

Abnormal liver function is acceptable.

Biliary obstruction for which a shunt has been placed is acceptable provided the shunt is in place for at least 10 days prior to the first dose of oxaliplatin to allow the liver function tests to stabilize.

No evidence of clinically significant neuropathy.

Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Breastfeeding should be discontinued if the mother is treated with oxaliplatin.

Must be able to understand and willing to sign a written informed consent document.

No chemotherapy or radiotherapy within 4 weeks prior to entering the study and no platinum therapy within 6 weeks prior to entering the study.

Not undergoing therapy with other investigational agents.

No known brain metastases.

No history of allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy.

No uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, or unstable angina pectoris, or cardiac arrhythmia.

No HIV-positive patients receiving anti-retroviral therapy (HAART).

No known allergy to erythromycin or indocyanine green.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2000-07; Study Completion 2001-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kraker AJ, Moore CW. Accumulation of cis-diamminedichloroplatinum(II) and platinum analogues by platinum-resistant murine leukemia cells in vitro. Cancer Res. 1988 Jan 1;48(1):9-13. PMID 3335002
- [Background] Pendyala L, Creaven PJ. In vitro cytotoxicity, protein binding, red blood cell partitioning, and biotransformation of oxaliplatin. Cancer Res. 1993 Dec 15;53(24):5970-6. PMID 8261411
- [Background] Rixe O, Ortuzar W, Alvarez M, Parker R, Reed E, Paull K, Fojo T. Oxaliplatin, tetraplatin, cisplatin, and carboplatin: spectrum of activity in drug-resistant cell lines and in the cell lines of the National Cancer Institute's Anticancer Drug Screen panel. Biochem Pharmacol. 1996 Dec 24;52(12):1855-65. doi: 10.1016/s0006-2952(97)81490-6. PMID 8951344